CLINICAL TRIAL: NCT01669161
Title: A Proof-of-Concept Pilot Study Assessing Vagus Nerve Stimulation (VNS) Paired With Rehabilitation for Improved Upper Limb Function After Stroke (MicroTransponder's Vivistim System)
Brief Title: Paired Vagus Nerve Stimulation (VNS) With Rehabilitation for Upper Limb Function Improvement After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroTransponder Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mt-St-01
Record Dates: First submitted 2012-08-15; First posted 2012-08-20 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
Keywords: Upper; Limb; Deficits; Rehabilitation; VNS
MeSH Terms: conditions — Stroke | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VNS (Experimental): VNS (vagus nerve stimulation) paired with rehabilitation as provided by the Vivistim System.
  Interventions: Device: Vivistim System
- Rehab Only (Active Comparator): Rehabilitation only (no implant, no VNS)
  Interventions: Other: Rehab Only

INTERVENTIONS:
Device: Vivistim System — The Vivistim System provides vagus nerve stimulation (VNS) with rehabilitation movements.
  Other Names: VNS, vagus nerve stimulation, paired VNS
  Arms: VNS
Other: Rehab Only — Rehabilitation without device implant and VNS
  Arms: Rehab Only

SUMMARY:
Patients (UK only) at least 6 months post stroke, with upper limb deficits, may enroll. Patients will be randomized to one of two groups - a group implanted with a device that allows pairing VNS with rehabilitation and a group that only receives rehabilitation (no implant). Patients have two baseline evaluations, one evaluation after implant but before initiation of treatment, and then six weeks of rehabilitation or rehabilitation + VNS, followed by post acute therapy evaluations at 1, 7, and 30 days after the 6-weeks of treatment. The intent is to assess safety and provide preliminary effectiveness information for VNS for upper limb functional improvement after stroke. Implanted patients may receive longer-term treatment and follow-up after the acute study.

ELIGIBILITY:
Major Inclusion Criteria:

1. History of unilateral supratentorial ischemic stroke that occurred at least 6 months prior
2. Age > 18 years and < 80 years
3. Right or left sided weakness of upper extremity

Major Exclusion Criteria:

1. Hemorrhagic stroke
2. Any deficits in language or attention that interferes with reasonable study participation
3. Presence of significant apraxia
4. Profound Sensory loss
5. Active major neurological or psychiatric diagnosis that would likely interfere with study protocol including alcohol or drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety | 6-weeks
  Assessment of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Dawson, MD, Principal Investigator — U. Glasgow
Locations (1):
- U. Glasgow / Western Infirmary, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dawson J, Pierce D, Dixit A, Kimberley TJ, Robertson M, Tarver B, Hilmi O, McLean J, Forbes K, Kilgard MP, Rennaker RL, Cramer SC, Walters M, Engineer N. Safety, Feasibility, and Efficacy of Vagus Nerve Stimulation Paired With Upper-Limb Rehabilitation After Ischemic Stroke. Stroke. 2016 Jan;47(1):143-50. doi: 10.1161/STROKEAHA.115.010477. Epub 2015 Dec 8. PMID 26645257
- See also: Abstract presented at the International Stroke Conference (ISC) — http://my.americanheart.org/idc/groups/ahamah-public/@wcm/@sop/@scon/documents/downloadable/ucm_471670.pdf